CLINICAL TRIAL: NCT02933931
Title: Long-term Immune Durability After Vaccination With the Vesicular Stomatitis Virus-vectored Zaire Ebola Candidate Vaccine (VSV-EBOV): a Prospective Observational Cohort Study
Brief Title: Immune Durability After VSV-EBOV Vaccination
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Siegrist Claire-Anne, Professor, University Hospital, Geneva
Other Study IDs: 2016-00918
Record Dates: First submitted 2016-10-11; First posted 2016-10-14 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Immune Response; Vaccination; Durability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood (RNA preservation)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- vaccinated with 5 x 10E7 pfu VSV-ZEBOV: Volunteers vaccinated in 2014 or 2015 with 5 x 10E7 pfu VSV-ZEBOV
- vaccinated with 10E7 pfu VSV-ZEBOV: Volunteers vaccinated in 2014 or 2015 with 10E7 pfu VSV-ZEBOV
- vaccinated with 3 x 10E5 pfu VSV-ZEBOV: Volunteers vaccinated in 2014 or 2015 with 3 x 10E5 pfu VSV-ZEBOV

SUMMARY:
This prospective observational cohort study will follow the roughly 100 adults who received the VSV-ZEBOV vaccine in the Geneva phase 1 randomized controlled trial in 2014-2015 in order to determine their long-term (5-year) immune response to vaccination.

DETAILED DESCRIPTION:
Background: During the Ebola epidemic of 2014-5, there was no proven therapy or prevention available beyond horizontal infection control measures. After the Canadian government donated 800 vials of the vaccine candidate VSV-EBOV to World Health Organization (WHO), the University Hospitals of Geneva agreed to perform a WHO-coordinated phase I/II double-blind, placebo-controlled randomized trial to assess the candidate's safety and immunogenicity healthy adult volunteers. The doses of 10 E7 pfu and 5 x 10 E7 pfu were tested in 35 and 16 volunteers, respectively, before a safety-driven study hold in late 2014. At trial resumption in early 2015, the remaining volunteers (n=51) received 3 x 10 E5 pfu. Thirteen volunteers received placebo. Among vaccinees, early immune responses were impressive, even at the lowest dose of 3 x 10 E5 pfu, and persisted well up to 6 months (last time point assessed). The trial successfully ended 12 months after injection. This prospective observational study will assess immune durability in this group of vaccinees at yearly time points up to five years post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participated and was vaccinated with a single injection of VSV-EBOV at a dose of either 3 x 10E5 pfu, 10E7 pfu or 5 x 10E7 pfu in the Geneva phase I VSV-EBOV vaccine trial (NCT02287480).
* Able to provide written, informed consent for this observational study.

Exclusion Criteria:

* Received additional vaccination with VSV-EBOV at similar or differing doses.
* Was lost to follow-up in the Geneva phase I VSV-EBOV vaccine trial

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are adults who were vaccinated according to the protocol of the Geneva phase I VSV-EBOV vaccine trial (NCT02287480) and who are willing and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
EBOV-specific IgG antibody titers measured by ELISA | 5 years after vaccination

SECONDARY OUTCOMES:
EBOV-specific IgG antibody titers measured by ELISA | 2, 3, and 4 years after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Anne Siegrist, MD, Principal Investigator — University of Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agnandji ST, Huttner A, Zinser ME, Njuguna P, Dahlke C, Fernandes JF, Yerly S, Dayer JA, Kraehling V, Kasonta R, Adegnika AA, Altfeld M, Auderset F, Bache EB, Biedenkopf N, Borregaard S, Brosnahan JS, Burrow R, Combescure C, Desmeules J, Eickmann M, Fehling SK, Finckh A, Goncalves AR, Grobusch MP, Hooper J, Jambrecina A, Kabwende AL, Kaya G, Kimani D, Lell B, Lemaitre B, Lohse AW, Massinga-Loembe M, Matthey A, Mordmuller B, Nolting A, Ogwang C, Ramharter M, Schmidt-Chanasit J, Schmiedel S, Silvera P, Stahl FR, Staines HM, Strecker T, Stubbe HC, Tsofa B, Zaki S, Fast P, Moorthy V, Kaiser L, Krishna S, Becker S, Kieny MP, Bejon P, Kremsner PG, Addo MM, Siegrist CA. Phase 1 Trials of rVSV Ebola Vaccine in Africa and Europe. N Engl J Med. 2016 Apr 28;374(17):1647-60. doi: 10.1056/NEJMoa1502924. Epub 2015 Apr 1. PMID 25830326
- [Background] Huttner A, Dayer JA, Yerly S, Combescure C, Auderset F, Desmeules J, Eickmann M, Finckh A, Goncalves AR, Hooper JW, Kaya G, Krahling V, Kwilas S, Lemaitre B, Matthey A, Silvera P, Becker S, Fast PE, Moorthy V, Kieny MP, Kaiser L, Siegrist CA; VSV-Ebola Consortium. The effect of dose on the safety and immunogenicity of the VSV Ebola candidate vaccine: a randomised double-blind, placebo-controlled phase 1/2 trial. Lancet Infect Dis. 2015 Oct;15(10):1156-1166. doi: 10.1016/S1473-3099(15)00154-1. Epub 2015 Aug 4. PMID 26248510
- [Derived] Huttner A, Agnandji ST, Combescure C, Fernandes JF, Bache EB, Kabwende L, Ndungu FM, Brosnahan J, Monath TP, Lemaitre B, Grillet S, Botto M, Engler O, Portmann J, Siegrist D, Bejon P, Silvera P, Kremsner P, Siegrist CA; VEBCON; VSV-EBOVAC; VSV-EBOPLUS Consortia. Determinants of antibody persistence across doses and continents after single-dose rVSV-ZEBOV vaccination for Ebola virus disease: an observational cohort study. Lancet Infect Dis. 2018 Jul;18(7):738-748. doi: 10.1016/S1473-3099(18)30165-8. Epub 2018 Apr 5. PMID 29627147